CLINICAL TRIAL: NCT06866093
Title: Evaluation of the Long-term Effect of Integrated Lifestyle Treatments on Dietary Habits, Sedentary Behavior, Anthropometry, Quality of Life in Female Breast Cancer Survivors, Through Traditional and Innovative Statistical Methods.
Brief Title: The Study is Observational and Retrospective: Lifestyle, BMI and Activity Physical.
Acronym: Lifestyle
Status: Active, not recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Principal Investigator, Livia S Augustin, Nutrition Researcher, PhD S.C. Epidemiologia e Biostatistica, National Cancer Institute, Naples
Other Study IDs: 44/22
Record Dates: First submitted 2025-02-19; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Body Weight Change
Keywords: Lifestyle study
MeSH Terms: conditions — Breast Neoplasms; Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — An exploratory secondary objective of the study, in a subset of the sample (N=40), includes an investigation of the microbiome of the breast tissue extracted during breast cancer surgery. This analysis is useful to determine breast cancer tissue microbiome and potential associations with different lifestyle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lifestyle: The cohort incluedes women (N=428) with a 5-year primary diagnosis of breast cancer eligible to participate in a diet and exercise trial (DEDiCa) in the previous years. Half of them actively participated in the trial and half did not for reasons other than health related issues. Those who consent to participate to the current observational study completed a series of questionnaires.
  Interventions: Other: Lifestyle

INTERVENTIONS:
Other: Lifestyle — Participants are asked to answer online survey questions about their anthropomethry, clinical conditions, socio-economical status, dietary habits, physical activity levels, quality of life, sleep quality and pshycological distress.

SUMMARY:
The goal of this observational-retrospective study is to learn about the long-term effects of a lifestyle intervention inclusive of dietary counselling and physical activity advice, on body weight in female breast cancer survivors who took the intervention in previous years compared to those who did not take it.

The main question it aims to answer is:

Does a long-term lifestyle intervention help to control body weight 5 years after breast cancer diagnosis? Participants are asked to answer online survey questions about their anthropomethry, clinical conditions, socio-economical status, dietary habits, physical activity levels, quality of life, sleep quality and pshycological distress.

DETAILED DESCRIPTION:
Investigators will use data from 428 women with a 5-yr primary diagnosis of BC (stages I-III at ages ≥30 <75 anni). Half of this sample (N=214) who followed integrated lifestyle treatment of behavioral modification of diet and physical activity conducted by Pascale Institute since 2016; the other half (N=214) will be patients who were eligible to participate but did not for logistic reasons.

The present study aims to enroll 428 women with prior primary diagnosis of breast cancer. Half of the patients (N = 214) had previously followed the lifestyle treatment of DEDiCa trial on the modification of eating and physical activity habits (Eudract n. 2015-005147-14) conducted by the Oncologic Institute Pascale in Naples (Italy) since Nov 2016; the other half of the patients were 214 who had refused to participate in the aforementioned trial for reasons unrelated to serious health conditions or progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Surgery for primary breast cancer performed at least 5 years prior to the interview.
2. Women who have joined the DEDiCa trial or who have refused to participate for reasons not related to serious health conditions or disease progression.
3. Those who are able to sign the informed consent.

Exclusion Criteria:

1. Age <30 years.
2. Primary diagnosis of metastatic breast cancer.
3. Diagnosis of other malignancies prior to the diagnosis of breast cancer.
4. Those who are unable to sign the informed consent or who deny to be contacted by telephone.

Ages: 30 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with a 5-year diagnosis of breast cancer, living in Italy and followed up in the participating hospitals.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of body weight in kilograms | Baseline
  The primary objective of the study is to evaluate whether an integrated lifestyle cancer treatment (L-INT) with nutritional and physical activity counseling, within the first year of diagnosis of histologically confirmed primary breast cancer, can result in better control of body weight (measured as BMI classes) after 5 years from diagnosis compared to those who had not adhered to integrated lifestyle treatments (no-INT).
Measurement of body height in meters | Baseline
  The primary objective of the study is to evaluate whether an integrated lifestyle cancer treatment (L-INT) with nutritional and physical activity counseling, within the first year of diagnosis of histologically confirmed primary breast cancer, can result in better control of body weight (measured as BMI classes) after 5 years from diagnosis compared to those who had not adhered to integrated lifestyle treatments (no-INT).

SECONDARY OUTCOMES:
Units on a Scale adherence to the Mediterranean diet. | Baseline
  The secondary objectives aim to evaluate the current adherence to the Mediterranean diet and the following variables: disease-free survival, new onset of chronic diseases (second cancer, diabetes, cardiovascular events, osteoporosis/bone fractures), quality of life including psychological distress and sleep quality. As an exploratory secondary objective, on a subgroup (N = 40), plans to study the microbiome of breast cancer tissue stored in the biobank of the Pascale Institute, to relate it to the characteristics of the disease and the patients' lifestyle.
Units on a Scale moderate physical activity. | Baseline
  The secondary objectives of study is moderate physical activity, together at the association between current adherence to the Mediterranean diet and the following variables: current body weight (BMI), disease-free survival, new onset of chronic diseases (second cancer, diabetes, cardiovascular events, osteoporosis/bone fractures), quality of life including psychological distress, quality of sleep and economic sustainability of the disease.
Units on a Scale the microbiome of breast tissue | Baseline
  As a secondary exploratory and innovative objective, on a subgroup (N=40), we plan to study the microbiome of the breast tissue stored in the biobank of the Pascale Institute, to relate it to the characteristics of the disease and the patient.
Units on a Scale of questionnaries quality of life | Baseline
  The study aim on quality of life including psychological distress, quality of sleep and economic sustainability of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Cancer Institute Foundation G. Pascale of Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: No